CLINICAL TRIAL: NCT05959473
Title: Idylla™ EGFR_IUO/3.20 Mutation Test a Clinical Trial Assay in the AstraZeneca Phase III NeoADAURA Clinical Trial (D516AC00001) Clinical Study Protocol
Brief Title: EGFR_IUO 3.20 Clinical Study Protocol
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants with FNA samples were enrolled
Sponsor: Biocartis NV (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BC-020066
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: NSCLC

STUDY DESIGN:
Masking Description: Specimens from NSCLC patient with FFPE FNA samples, will be extracted and tested with the Idylla EGFR_IUO/3.20.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Idylla EGFR_IUO/3.20 Mutation Test — Clinical Performance Study Protocol for Idylla EGFR_IUO/3.20 Mutation Test The EGFR_IUO/3.20 is automated on the Idylla™ Platform, which executes the entire process from sample to result including sample liquefaction, cell lysis, real-time PCR amplification/detection, and data analysis and reporting.

SUMMARY:
An interventional, prospective clinical performance study protocol, for the testing of DNA extracted from FFPE Fine needle aspirate samples, using the Idylla EGFR_IUO/3.20, from patients with Non-Small Cell Lung Cancer screened in AstraZeneca's NeoADAURA clinical trial (Protocol No. D516AC00001)

DETAILED DESCRIPTION:
This is a prospective, interventional diagnostic study using the For Investigational Use Only EGFR_IUO/3.20 for FFPE FNA sections. Screened patients with available FNA specimens, collected per SoC, who are found to have exon 19 deletions or L858R mutations in the EGFR gene based on the results of EGFR_IUO/3.20 and who meet all other study eligibility criteria will be randomized into one of three arms of the NeoADAURA study: neoadjuvant osimertinib as monotherapy or in combination with pemetrexed/platinum chemotherapy, versus pemetrexed/platinum chemotherapy plus placebo.

The use of the investigational IVD does not require invasive sampling that is not part of standard of care (SoC). Investigational testing for patient selection will be performed on FFPE FNA specimens, obtained as SoC for diagnosis and/or pathologic staging prior to definitive surgery. By using available specimens obtained as SoC, there is no risk to patients as a result of invasive sampling for EGFR testing.

ELIGIBILITY:
Inclusion Criteria:

• All patients who provided consent (by signing and dating the Consent Form for AstraZeneca NeoADAURA Protocol No. D516AC00001), may be included in the device study.

Exclusion Criteria:

* Patients whose FFPE FNA samples are not Clinical Trial Assay evaluable will be excluded from the study.
* Patients with samples identified for the study which have insufficient testing material will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 7 business days
  EGFR_IUO/3.20 as a screening test in Phase 3 of clinical trial (Protocol D516AC00001), in order to identify patients (with NSCLC) with EGFR mutation positive (Exon 19 deletion and/or L858R) for inclusion in study (D516AC00001)